CLINICAL TRIAL: NCT02786459
Title: Detection and Localization of Carcinoma Using High Resolution Transrectal Imaging - Proof of Concept Study
Acronym: ProxiScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hybridyne Imaging Technologies Inc (Unknown); Aytu BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-8723-C
Record Dates: First submitted 2016-05-04; First posted 2016-06-01 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: Prostate; Local Recurrence; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging; Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Post Radical Prostatectomy (Experimental): Up to n=30 evaluable male patients, between ages 30-75, who were previously diagnosed with PCa, have undergone a RP at least 6 months before imaging and who experience rising PSA (biochemical failure). The RP group (n=30) will be stratified into PSA subgroups <0.005, 0.005-<0.2, >0.2.
  Intervention: men will be imaged with ProxiScan, SPECT-CT and MRI.
  Interventions: Device: ProxiScan; Device: Magnetic Resonance Imaging; Device: SPECT-CT
- Active Surveillance (Active Comparator): Up to n=10 men, between ages 30-75, on active surveillance with known prostate adenocarcinoma diagnosis and multiple positive biopsies.
  Intervention: men will be imaged with ProxiScan, SPECT-CT and MRI, and also undergo a TRUS biopsy.
  Interventions: Device: ProxiScan; Device: Magnetic Resonance Imaging; Device: SPECT-CT
- Multiple Negative Biopsies (Experimental): Up to n=20 men, between ages 30-75, who have previously undergone one/or multiple negative biopsies, with elevated PSA (≥4 ng/mL) and/or an abnormal digital rectal exam suspicious for prostate cancer with a planned sextant prostate biopsy but who do not have a definitive PCa diagnosis.
  Intervention: men will be imaged with ProxiScan, SPECT-CT and MRI, and also undergo a TRUS biopsy.
  Interventions: Device: ProxiScan; Device: Magnetic Resonance Imaging; Device: SPECT-CT

INTERVENTIONS:
Device: ProxiScan — ProxiScan probe will be coupled with ProstaScint (a radioactive tracer) and used to perform imaging to detect small lesions in the pelvis that will otherwise be hard to detect with conventional imaging modalities.
Device: Magnetic Resonance Imaging — Used as a comparative to ProxiScan.
Device: SPECT-CT — Used as a comparative to ProxiScan.

SUMMARY:
An exploratory, feasibility and proof-of-concept study to evaluate the capability of a rectal probe scintigraphy device (ProxiScanTM) to detect PSMA specific radiopharmaceutical agent (ProstaScintÂ®; as a surrogate marker for prostate cancer) in patients who have undergone a radical prostatectomy for their disease, patients with multiple negative prostate biopsies and patients with known primary prostate cancer. Developed by Hybridyne Imaging Technologies, Inc. ProxiScanTM is a small cadmium zinc telluride (CST)-based compact gamma camera. It is the same size as a trans-rectal ultrasound (TRUS), currently used for prostate biopsy guidance. Men with multiple positive biopsies will be considered controls. Prostate cancer sextant biopsy histology results will be correlated with ProxiScanTM, TRUS, MRI and SPECT/CT. The investigators hypothesize that it will be safe and feasible to utilize a rectal probe scintigraphy (ProxiScanTM) to detect PSMA specific ProstaScintÂ®, thus identifying and localizing the tumour sites within the prostate and surrounding areas.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Rising PSA (biochemical failure) following radical prostatectomy. Group 2: Rising PSA (>10ng/ml) and/or abnormal digital rectal exam suspicious for prostate cancer. Previously negative prostate biopsies.

Group 3: Scheduled biopsy for known PCa (patient on AS). At least 1 previously positive prostate biopsy for adenocarcinoma of the prostate.

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Sufficient time period to complete the imaging protocol and 7 to 9 day safety follow-up assessment without therapeutic intervention.
* Patient is judged by the Investigator to have the initiative and means to provide written consent and be compliant with the protocol and be able and commits to make the required study visits.
* Ambulatory with ECOG performance status of 0 or 1 (see appendix section).
* Patient is between 35 and 75 years of age.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

* Patient or physician plans definitive concomitant chemotherapy, therapeutic radiation treatment, biologic treatment and/or local ablative treatment for cancer within the interval of study participation.
* Patients with pacemakers, neurostimulators, and foreign metal bodies will be excluded as they will be unable to undergo an MRI and SPECT-CT.
* Prior history of murine antibody infusion, patients who are hypersensitive to products of murine origin or indium-111 chloride.
* Prior therapeutic pelvic irradiation.
* Recent prostate biopsy, within 1 month of study enrollment.
* Patient with contraindications to TRUS-guided prostate biopsy (continuous need for anti-coagulation, no rectum, etc.)
* Clinical evidence of prostatitis, or other benign prostate gland abnormality, that would explain elevated PSA and/or (digital rectal exam) DRE findings.
* Active malignancy or therapy for malignancy within 6 months, other than basal or squamous cell carcinoma of the skin.
* Patient received a radiopharmaceutical which was within 5 physical half-lives at the time of study imaging.
* Severe psychiatric or medical illness that may interfere with compliance with the study protocol or follow-up as deemed by the investigator.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Tumor localization. | Within 2 days of imaging.
  Identification of tumour and/or tumour recurrence in the pelvis with imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided